CLINICAL TRIAL: NCT06199895
Title: Clinical Efficacy and Safety of Paclitaxel Polymeric Micelles for Injection in the Treatment of Patients With Taxanes-resistant Pancreatic Adenocarcinoma, Cholangiocarcinoma, Lung Cancer, Gastric Cancer, Esophageal Carcinoma, or Breast Cancer
Brief Title: Clinical Efficacy and Safety of Paclitaxel Polymeric Micelles for Injection in the Treatment of Patients With Taxans-resistant Pancreatic Adenocarcinoma, Cholangiocarcinoma, Lung Cancer, Gastric Cancer, Esophageal Carcinoma, or Breast Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Liu Huang (Other)
Responsible Party: Sponsor-Investigator, Liu Huang, Professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PM1
Record Dates: First submitted 2023-12-29; First posted 2024-01-10 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Pancreatic Adenocarcinoma; Cholangiocarcinoma; Lung Cancer; Stomach Cancer; Esophageal Carcinoma; Breast Cancer
MeSH Terms: conditions — Cholangiocarcinoma; Lung Neoplasms; Stomach Neoplasms; Esophageal Neoplasms; Breast Neoplasms | interventions — Injections

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Paclitaxel Polymeric Micelles for Injection (Experimental): Subjects are given paclitaxel polymeric micelles for injection, three weeks constitutes one cycle of treatment.
  Interventions: Drug: Paclitaxel Polymeric Micelles for Injection

INTERVENTIONS:
Drug: Paclitaxel Polymeric Micelles for Injection — 300mg/m2 of Paclitaxel Polymeric Micelles for Injection is intravenously administrated for ≥ 3 hours without special infusion device. The frequency of administration is once every 3 weeks (Q3W), and 3 weeks constitutes a treatment cycle.

SUMMARY:
This study is a single-center, single-arm, open-label, phase II clinical trial designed to evaluate the efficacy and safety of Paclitaxel Polymeric Micelles for Injection for the treatment of patients with advanced pancreatic adenocarcinoma, cholangiocarcinoma, lung cancer, gastric cancer, esophageal carcinoma, or breast cancer that are resistant to Taxanes.

Subjects are given paclitaxel polymeric micelles for injection, three weeks constitutes one cycle of treatment.

If subject does not develop disease progression , the subject continues treatment until disease progression (RECIST 1.1) or develops an intolerable toxicity, initiation of a new anti-cancer drug, withdrawal from the study, death, or loss of follow-up.

This is a single-arm, small-sample clinical study with the primary efficacy goal of objective remission rate (ORR). The parameters of the trial were set: assuming a class I error of 0.025 unilaterally, power=90%, and a 15% improvement in ORR for objective remission rate, a total of 20 subjects would be required, and a total of 25 would be required for enrolment, taking into account a 20% shedding.

ELIGIBILITY:
Inclusion Criteria:

* 1.Male or female 18 years and older; 2.Patients with advanced pancreatic adenocarcinoma, cholangiocarcinoma, lung cancer, gastric cancer, esophageal carcinoma, or breast cancer diagnosed by histological or cytological pathology; must have an evaluable lesion; 3.Previous treatment regimen includes Taxanes and is resistant to Taxanes (including patients with initial failure to remit or progression after remission) or previous use of Taxanes for at least 2 cycles without tumour shrinkage and the patient is not satisfied with current stable efficacy and is willing to be enrolled in this study; 4.ECOG (Eastern Cooperative Oncology Group) score ≤ 2 points; 5.expected survival of at least 3 months; 6.Blood routine examination meets the following criteria:

  1. WBC≥3.0×109 /L，ANC≥1.5×109 /L;
  2. PLT≥100×109 /L；
  3. Hb≥80g/L； 7.Blood biochemical examination must meet the following criteria:

  <!-- -->

  1. Total bilirubin ≤1.5 times the upper limit of normal (ULN)；
  2. Aspartate aminotransferase (AST), alanine aminotransferase (ALT), or alkaline phosphatase (ALP) ≤2.5 times ULN (ALT, AST, or ALP≤ 5×ULN for subjects with liver metastases, and ALP≤10×ULN for subjects with bone metastases);
  3. Creatinine clearance (calculated using Cockcroft-Gault formula) ≥50 ml/min； 8.Functions of major organs such as heart, lung, liver and kidney are basically normal； 9.Subjects have good compliance and voluntarily comply with the clinical trial protocol during the study, followed up by the investigators； 10.All women of childbearing age, men of childbearing potential, or their spouses who have no plans to have children or donate sperm during the entire trial period and up to 6 months after the last dose of medication, or who voluntarily used effective contraception; Women of childbearing age who have a negative blood/urine pregnancy test within 7 days prior to enrollment； 11.Subjects had fully understood the study and voluntarily signed the informed consent form .

Exclusion Criteria:

* 1.Subjects with an allergic history to experimental drugs or any excipients； 2.Subjects with acute or chronic infections that have not been eliminated, or subjects with other serious diseases at the same time; 3.Subjects with active hepatitis and uncontrolled by antiviral therapy, or liver metastasis is more than 3/4 of the whole liver； 4.Subjects with third-space effusions (e.g., moderate-to-massive pleural effusion, moderate-to-massive pericardial effusion, ascites) that cannot be controlled by drainage or other means; 5.Subjects with mental illness or disorder, poor compliance, or inability to cooperate, or describe treatment responses； 6.Subjects who cannot tolerate chemotherapy due to severe organic disease or major organ failure, such as decompensated heart and lung failure； 7.Subjects with bleeding disorders； 8.Subjects with organ transplant; 9.Subjects with bad drug addicts, long-term alcoholics, infectious diseases such as AIDS； 10.Subjects who still have grade ≥2 toxicity from previous antineoplastic therapy (except alopecia and grade ≤2 neurotoxicity caused by platinum) at enrollment; 11.Subjects are considered not able to complete the trial or otherwise unfit to participate in the study by the investigators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2023-11-28 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | Baseline to measured PD（up to 24 months)
  Proportion of subjects who have achieved complete response (CR) or partial response (PR) (RECIST 1.1)

SECONDARY OUTCOMES:
Progression-Free-Survival | Randomization to measured PD or date of death from any cause（up to 24 months)]
  PFS(Progression-Free-Survival) was the time from randomization until the date of objectively determined progressive disease (PD) or death due to any cause, whichever occurred first.
Disease Control Rate | Baseline to measured PD（up to 24 months)
  Proportion of subjects who have achieved complete response (CR), partial response (PR) or stable disease (SD) (RECIST 1.1)
Overall Survival | Randomization to date of death from any cause（up to 24 months)]
  The time from randomization to death.
Incidence of adverse events | up to 24 months
  Safety

CONTACTS AND LOCATIONS:
Overall Officials: Xianglin Yuan, Principal Investigator — Tongji Hospital
Locations (1):
- Tongji Hospital, Wuhan, Hubei, China